CLINICAL TRIAL: NCT03978910
Title: Rendering of a Local 1g Environment for Enhanced Motor Learning in Altered Gravity
Acronym: Sim1g
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-210
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weigthlessness (Experimental): during a flight
  Interventions: Other: measurements of the accuracy of the reaching movements

INTERVENTIONS:
Other: measurements of the accuracy of the reaching movements — Euclidian distance between final position and target

SUMMARY:
Human motor adaptation is crucial to adapt to new environments, such as altered gravity. Dexterous manipulation and fine movements in space require learning new coordinated motor actions. Traditionally, adaptation mechanisms have been tested in laboratories with robotic devices that perturb specific task parameters unbeknownst to the participant. Over repetition, participants build a more accurate representation of the task dynamics and, eventually, improve performance. These perturbations are applied locally on the hand or limb while the dynamics of the rest of the body remains unaltered. These approaches are therefore limitative since they do not reflect ecological adaptation to globally changed dynamics, such as new gravitational environments. Parabolic flights, centrifuges and water immersion allow circumventing these limitations. Previous investigations in these contexts have highlighted the role of the global context in motor adaptation. However, it is unknown if global learning could benefit from exploiting known local dynamics. Here, we design an original task that will capture both the learning of arm movement kinematics as well as grasping forces for object manipulation in an ecologically valid design. We test whether executing this task in hypogravity with rendering of Earth gravity locally at the hand is beneficial or detrimental to task performance. By adopting the "negative picture" of conventional robotic approaches, these results will further our understanding of basic motor adaptation and provide insightful information on the optimal design and control of human-machine interfaces and wearable robots in space environments and other immersive dynamics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women).
* Aged from 18 to 65.
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC).
* Who accepted to take part in the study.
* Who can take scopolamine or nautamine (medication against airsickness).
* Who have given their informed written stated consent.
* Who have passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination) and have been declared fit to fly. The examination must be less than one year before the experiment flight. There will be no additional test performed for participant selection.

Exclusion Criteria:

* Persons who took part in a previous biomedical research protocol, of which exclusion period is not terminated.
* Persons with any history of cerebral, cardiovascular or vestibular diseases.
* Persons with history of psychiatric diseases, including anxiety disorder.
* Persons whose medical condition has changed since the class 2-like medical examination.
* Pregnant women (urine pregnancy test for women of childbearing potential).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
accuracy of the reaching movements | baseline
  Euclidian distance between final position and target

CONTACTS AND LOCATIONS:
Locations (1):
- Caen Univerity Hospital, Caen, France